CLINICAL TRIAL: NCT07201753
Title: Exploring the Relationship Between Hospital-integrated Care Services and Caregiver Burden at a Medical Center in Northern Taiwan.
Brief Title: Hospital-integrated Care Services
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202506121RINB
Record Dates: First submitted 2025-08-14; First posted 2025-10-01 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Caregiver Burden of Caregivers; Hospital-Integrated Care Services

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore the relationship between hospital-integrated care services and caregivers' psychological outcomes. The study will be conducted as a cross-sectional observational design at a medical center in northern Taiwan. Data will be collected from primary caregivers of hospitalized patients through validated questionnaires. The findings are expected to provide insights into improving caregiver support and enhancing patient and caregiver experiences during hospital stays.

ELIGIBILITY:
Inclusion Criteria:

* Participants include inpatients receiving integrated inpatient care services at our hospital and their primary family caregivers. The patient or family member must have signed the consent form for integrated inpatient care services. The specific conditions are as follows:

  1. Primary Caregiver Criteria:

  <!-- -->

  1. The primary caregiver is a family member aged 18 years or older who can communicate in Mandarin or Taiwanese.
  2. The family member is willing to sign the participant consent form. 2.Patient Criteria:

  <!-- -->

  1. The patient has been admitted to the pilot ward for at least 24 hours.

Exclusion Criteria:

1. Patients who are discharged or transferred out of the pilot ward within 24 hours of admission.
2. If a patient is re-hospitalized during the study enrollment period and their primary caregiver is the same as in the previous enrollment, the subsequent duplicate case will be excluded.
3. Patients without family members will be enrolled in the ward's mandatory integrated inpatient care service program, but follow-up care issues will be handled by social workers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary caregivers of hospitalized adult patients receiving integrated inpatient care services at a medical center in northern Taiwan. Caregivers must be aged 18 years or older and able to complete the study questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Total score of caregiver burden as measured by the Zarit Burden Interview (ZBI-22) | Within 48 hours prior to hospital discharge.
  The Traditional Chinese version of the ZBI-22 includes 22 Likert-type items (0-4); total scores range from 0 to 88, with higher scores indicating greater burden.

SECONDARY OUTCOMES:
Total score of caregiver burden as measured by the Caregiver Burden Inventory (CBI) | Within 48 hours prior to hospital discharge.
  The Traditional Chinese version of the CBI includes 24 Likert-type items (0-4); total scores range from 0 to 96, with higher scores indicating greater burden across multiple domains.
Subscale scores of anxiety and depression as measured by the Hospital Anxiety and Depression Scale (HADS) | Within 48 hours prior to hospital discharge.
  The Traditional Chinese version of HADS contains 14 items, 7 for anxiety and 7 for depression. Each item is scored 0-3; subscale scores range from 0 to 21, with higher scores indicating more severe symptoms.
Domain mean scores of inpatient satisfaction as measured by the standardized hospital inpatient satisfaction survey | Within 48 hours prior to hospital discharge.
  The hospital's standardized inpatient satisfaction survey includes 31 items. Each item is rated on a 5-point Likert-type scale, with response anchors varying by question (e.g., from "very sufficient" to "very insufficient," or from "strongly agree" to "strongly disagree"). Scores are calculated as domain means, with higher scores indicating greater inpatient satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei City, Taiwan